CLINICAL TRIAL: NCT02182544
Title: Phase III Double-blind Comparative Study of WAL801CL Dry Syrup in Paediatric Perennial Allergic Rhinitis
Brief Title: WAL801CL (Epinastine Hydrochloride) Dry Syrup in Paediatric Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 262.258
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

ARMS (2):
- WAL801CL dry syrup + Placebo (Experimental)
  Interventions: Drug: WAL801CL dry syrup; Drug: Ketotifen fumarate dry syrup placebo
- Ketotifen fumarate dry syrup + Placebo (Active Comparator)
  Interventions: Drug: Ketotifen fumarate dry syrup; Drug: WAL 801 CL dry syrup placebo

INTERVENTIONS:
Drug: WAL801CL dry syrup
  Arms: WAL801CL dry syrup + Placebo
Drug: Ketotifen fumarate dry syrup
  Arms: Ketotifen fumarate dry syrup + Placebo
Drug: Ketotifen fumarate dry syrup placebo
  Arms: WAL801CL dry syrup + Placebo
Drug: WAL 801 CL dry syrup placebo
  Arms: Ketotifen fumarate dry syrup + Placebo

SUMMARY:
Study to investigate the efficacy of WAL801CL Dry Syrup in comparison with ketotifen fumarate on pediatric perennial allergic rhinitis and to evaluate the safety of WAL801CL Dry Syrup compared to ketotifen fumarate and to confirm the appropriateness of dosage of WAL801 Dry Syrup.

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age or younger
* Body weight of 14 kg or more
* Typical symptoms of perennial allergic rhinitis, and within 2 or higher score of serum specific immunoglobulin E (IgE) caused by house dust (HD) or mite in the data obtained with the past one year
* "Moderate" or "Severe" in the Allergic Rhinitis Severity Classification during the observation period
* The Patient Diary can be entered by the patient or parent
* Outpatients

Exclusion Criteria:

* Absolute necessity of treatment with a drug that may affect the evaluation of the effect of the investigational drug (e.g., anti-histamines, anti-allergics, steroid, vasopressors). Patients being treated with the following drugs, however, may be included

  * Intal® Oral or Inhalation
  * Any eye drops other than Zaditen® Eye Drop
  * External preparations (liniment, poultice)
* Initiation of desensitisation therapy within the past 6 months
* Onset of acute upper respiratory inflammation during the observation period
* Nasal disease, such as acute or chronic rhinitis, nasal polyp, hypertrophic rhinitis, septal deviation*, sinusitis*, and hypertrophied adenoid*, of such a degree that the disease affects evaluation of the effect of the test drug (*: X-ray examination will be conducted if necessary)
* That pollen (cider, ragweed, Japanese cypress, orchard grass, etc.) is a double antigen, and that the study will be conducted in the season of air-borne pollen, and symptoms may be exacerbated by pollen
* Present or past history of a convulsive disease, such as epilepsy (convulsion threshold values may be decreased by the comparator drug, ketotifen fumarate)
* Clinically significant abnormal changes in laboratory measurements, and thus judgement that the patient is ineligible for inclusion in this study; however, if the patient is judged as falling into Grade 2 or more according to the MHW (Ministry of health and welfare) Adverse Reaction Severity Classification Criteria, the patient will be excluded from the study
* Clinically significant renal, hepatic or cardiac disease, or other complications, and thus judgement that the patient is ineligible for inclusion in the study; however, if the patient is judged as falling into Grade 2 or more according to the MHW Adverse Reaction Severity Classification Criteria, the patient will be excluded from the study
* Past history of drug allergy
* 1 month, or 6 times as long as the half life of the investigational drug if it is over 1 month, will not have passed since participation in any other clinical trial study, at the time of the initiation of this study
* Judgement by the Principal Investigator or Investigator that the patient is ineligible for inclusion in this study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2001-06; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Total severity scores of nasal symptoms judged by the physician | 2 weeks of first administration of study drug

SECONDARY OUTCOMES:
Severity score for each nasal symptom given by the physician | 2 weeks of first administration of study drug
Nasal symptom score in the diary | 2 weeks
Total scores for nasal symptoms in the diary | 2 weeks of first administration of study drug
Severity score for allergic rhinitis according to the Allergic Rhinitis Severity Classification | 2 weeks
Impression of the patient or the parent | week 2 after first administration of study drug
Occurrence of adverse events | up to 2 weeks after administration of study drug
Number of patients with abnormal changes from baseline in laboratory tests (hematology, biochemistry, urinalysis) | Baseline and week 2